CLINICAL TRIAL: NCT01351285
Title: Comparison of Effect-site Concentration of Remifentanil for Preventing Cough Against Endotracheal Tube During Anesthetic Emergence According to Anesthetics (Sevoflurane, Desflurane, and Propofol)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 4-2011-0019
Record Dates: First submitted 2011-05-04; First posted 2011-05-10 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Female Patients Undergoing Thyroidectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sevo group (Experimental): undergoing sevoflurane-remifentanil anesthesia
  Interventions: Drug: up-and-down method to find out effective concentration of remifentanil for preventing cough
- Des group (Active Comparator): undergoing desflurane-remifentanil anesthesia
  Interventions: Drug: up-and-down method to find out effective concentration of remifentanil for preventing cough
- Pro group (Active Comparator): undergoing propofol-remifentanil anesthesia
  Interventions: Drug: up-and-down method to find out effective concentration of remifentanil for preventing cough

INTERVENTIONS:
Drug: up-and-down method to find out effective concentration of remifentanil for preventing cough — During the emergence from anesthesia, if the patient did not cough, the extubation was defined as smooth emergence and the predetermined effect site concentration of remifentanil for the subsequent patient was decreased by 0.5 ng/mL. Likewise, if the patient coughed anytime around extubation, it was considered a failed smooth emergence and the predetermined effect site concentration for the next patient was increased by 0.5 ng/mL. This up-and-down method was conducted independently for each of the three groups. EC50 of the remifentanil of each group was obtained using the Dixon's method.

SUMMARY:
It has been reported that target-controlled infusion of remifentanil can reduce cough against endotracheal tube during emergence from general anesthesia. We hypothesized that effective concentration of remifentanil for preventing cough during anesthetic emergence varies depending on the type of main anesthetic agents which is administered with remifentanil during general anesthesia. The purpose of this study is to evaluate the effective concentrations of remifentanil to prevent coughing during emergence from general anesthesia according to main anesthetic agent (sevoflurane, desflurane, and propofol).

ELIGIBILITY:
Inclusion Criteria:

* aged 20-60
* ASA classification I~II
* female patients
* patients who undergoing thyroidectomy

Exclusion Criteria:

* Patients with acute or chronic respiratory disease
* patient who has smoking history
* patient who has hypertension
* patient who has esophageal reflux
* patient who having an expectorant or cough remedy

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2011-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
occurrence of cough | From the completion of surgery to 5minute after extubation
  We will assess the occurrence of cough during emergence from general anesthesia in female patients undergoing target controlled infusion of remifentanil at predetemined concentration.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Seoul, South Korea